CLINICAL TRIAL: NCT01040975
Title: Teen CHAT: Improving Physician Communication With Adolescents About Healthy Weight
Acronym: TeenCHAT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00016206; 1R01HL092403-01A2 (NIH)
Record Dates: First submitted 2009-12-29; First posted 2009-12-30 (Estimated); Last update posted 2016-09-23 (Estimated); Status verified 2016-09

CONDITIONS: Communication; Obesity; Nutrition; Physical Activity; Sleep
MeSH Terms: conditions — Communication; Obesity; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Motivational Interviewing intervention (Experimental): Web-based intervention targeting MD communication and Summary Report
  Interventions: Behavioral: Web-based intervention targeting MD communication; Summary Report
- Control (No Intervention): MD receives Summary Report only

INTERVENTIONS:
Behavioral: Web-based intervention targeting MD communication; Summary Report — Web-based intervention targeting MD communication; Summary Report detailing 6 risk factors for adolescent overweight/obesity developed by study team
  Other Names: Tailored Web-based intervention developed by study team; Tailored Summary Report
  Arms: Motivational Interviewing intervention

SUMMARY:
The purpose of this study is to teach primary care physicians effective ways to counsel overweight and obese adolescent patients to attain a healthy weight. Fifty physicians and up to 660 adolescent patients from Duke University Health System (DUHS) Primary Care Clinics will take part in this study.

Patients will be identified by research study staff and asked if they would be willing to have their clinic visit audio recorded for research purposes. There are three phases of data collection. First, baseline encounters (n=200, 4 per physician) are audio recorded. Then, half of the physicians will be randomized to receive a tailored web-based intervention containing information about evidence-based techniques to help adolescents attain a healthy weight. A new set of 200 encounters (4 per physician) will be audio recorded. Then, all physicians will receive a Summary Report that outlines the adolescent's high risk behaviors that contribute to weight (sweetened beverages, fast food, breakfast, physical activity, screen time, and sleep) and a new set of 200 encounters will be audio recorded.

Data will be collected by trained data technicians, in-person and over the phone. Data is collected on laptop computers and then downloaded into password protected electronic files on a secure network server. All participants (adolescent patients and physicians) will be assigned a code number that is the sole identifier on all study data forms. Prior to and after coding, digital files will be stored in password protected directories to which only the data technicians and project manager have access. The web-based intervention will be password protected.

ELIGIBILITY:
Inclusion Criteria for MDs:

* Specialty is Family Practice or Pediatrics
* Located in participating clinic
* Not planning to leave clinic in the next two years

Inclusion Criteria for teen patients:

* English-speaking
* BMI z-score >85th percentile
* age 12-18
* not pregnant
* have parental consent to participate if over 18
* have visit at least 7 days in the future
* have access to a telephone

Exclusion Criteria for teen patients:

* BMI z-score <85th percentile
* not English speaking
* pregnant
* <12 or older than 18
* incompetent for interview
* seen primarily by non-physician provider

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 684 (Actual)
Dates: Start 2009-09; Primary Completion 2013-12 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Physician communication | after CD-ROM phase

SECONDARY OUTCOMES:
Summary Report | After Summary Report Phase
  Assess whether summary report increases whether physicians address six health risk behaviors
Adolescent Nutrition, Physical Activity, and BMI Z-score | 3 months post-visit
  Examine whether patients whose MD was in the MI education arm improved their nutrition, physical activity, and BMI z-score 3 months post-visit more than patients whose MD was in the control arm.

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn I Pollak, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center - Cancer Prevention, Detection and Control, Durham, North Carolina, United States

REFERENCES:
- [Derived] Bodner ME, Lyna P, Ostbye T, Bravender T, Alexander SC, Tulsky JA, Lin PH, Pollak KI. Accuracy and congruence of physician and adolescent patient weight-related discussions: Teen CHAT (Communicating health: Analyzing talk). Patient Educ Couns. 2018 Dec;101(12):2105-2110. doi: 10.1016/j.pec.2018.07.022. Epub 2018 Jul 26. PMID 30115415
- [Derived] Pollak KI, Tulsky JA, Bravender T, Ostbye T, Lyna P, Dolor RJ, Coffman CJ, Bilheimer A, Lin PH, Farrell D, Bodner ME, Alexander SC. Teaching primary care physicians the 5 A's for discussing weight with overweight and obese adolescents. Patient Educ Couns. 2016 Oct;99(10):1620-5. doi: 10.1016/j.pec.2016.05.007. Epub 2016 May 9. PMID 27228899
- [Derived] Pollak KI, Coffman CJ, Tulsky JA, Alexander SC, Ostbye T, Farrell D, Lyna P, Dolor RJ, Bilheimer A, Lin PH, Bodner ME, Bravender TD. Teaching Physicians Motivational Interviewing for Discussing Weight With Overweight Adolescents. J Adolesc Health. 2016 Jul;59(1):96-103. doi: 10.1016/j.jadohealth.2016.03.026. Epub 2016 May 5. PMID 27155958
- [Derived] Ostbye T, Lyna P, Bodner ME, Alexander SC, Coffman C, Tulsky JA, Dolor R, Pollak K. The Effect of Parental Presence on Weight-Related Discussions Between Physicians and Their Overweight Adolescent Patients. Clin Pediatr (Phila). 2015 Oct;54(12):1218-20. doi: 10.1177/0009922814566027. Epub 2015 Jan 9. No abstract available. PMID 25575503
- [Derived] Alexander SC, Fortenberry JD, Pollak KI, Bravender T, Davis JK, Ostbye T, Tulsky JA, Dolor RJ, Shields CG. Sexuality talk during adolescent health maintenance visits. JAMA Pediatr. 2014 Feb;168(2):163-9. doi: 10.1001/jamapediatrics.2013.4338. PMID 24378686